CLINICAL TRIAL: NCT01050881
Title: Assessment of the Impact of Notification of Blood Donors Testing Positive for Microbiology Markers: What is the Psychological Impact of Notification and Does the Method of Notification Influence the Outcome?
Brief Title: Notification of Donors With Positive Microbiology Markers
Status: Completed | Type: Observational
Sponsor: NHS Blood and Transplant (Other Government)
Collaborators: Welsh Blood Service (Other); Scottish National Blood Transfusion Service (Unknown); Irish Blood Transfusion Service (Other)
Responsible Party: Sponsor
Other Study IDs: 001/DNS
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Human Immunodeficiency Virus; Hepatitis B; Hepatitis C; Human T-lymphotropic Virus I & II; Creutzfeldt-Jakob Syndrome
Keywords: blood donor notification; emotional response; variant Creutzfeldt-Jacob Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B; Hepatitis C; Creutzfeldt-Jakob Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Positive Blood Donors: Blood donors testing positive for HIV, HBV, HCV or HTLV in 2008 and 2009. Donors notified of increased risk of vCJD in 2005.

SUMMARY:
Each year around 200 blood donors in the UK are found to be infected with blood-borne diseases (HIV, hepatitis B, hepatitis C, and HTLV), while several others have been identified as having an increased risk of variant Creutzfeldt-Jakob Disease (vCJD). Although the notification procedures for these infections vary, their effectiveness and appropriateness have never been evaluated in a systematic study.

The proposed research has been designed to assess the responses of blood donors to notification and their satisfaction with how they were informed about the infection. The study will be implemented using standard questionnaire-based measures (French et al, 2004; Marteau & Bekker, 1992).

The study will involve approximately 600 blood donors who were informed of an infection or possible infection with blood-borne diseases in 2008 and 2009, and approximately 100 donors notified of possible risk of vCJD infection in 2005. A comparable group of 2005 donors will be included to control for the effects of time. As the majority of donors testing positive donated to NHS Blood and Transplant (NHSBT), the participants will be identified from the NHSBT database only, and their availability confirmed through their GP or specialist clinician. A standardized questionnaire will be then sent to all those identified as eligible.

The study will last 12 months, but direct participant involvement will be limited to the time required to complete the questionnaire, which should take under one hour. To safeguard confidentiality, no identifiable personal data will be used in the analysis. Where demographic or medical information already held by NHSBT is retrieved to minimise response burden, this will be pseudonymised before use.

The study is sponsored by the blood services for England, Wales, Scotland and Northern Ireland. The results will be used to inform notification procedures in the future.

DETAILED DESCRIPTION:
The purpose of the study is to assess the impact of notification of blood donors testing positive for microbiology markers for blood-borne and (mostly) currently incurable infections (hepatitis B, hepatitis C, HIV, HTLV and vCJD). Specifically, the study will focus on donors' responses to being notified of an infection or possible infection, and their satisfaction with the notification process. The data collected will be used to examine predictors of satisfaction and thus help inform notification procedures in the future.

In the UK, all donations are unpaid and voluntary, which is considered to be the safest method of blood collection (WHO Global Database on Blood Safety (GDBS) and Blood Safety Indicators). Out of the 1.9 million UK blood donations in 2008, only 187 (>0.01%) tested positive. With such low incidence and focus on blood safety, the deferred donor management is largely informed by anecdotal evidence and historical developments. The notification process is standardised within each blood service (e.g. NHSBT Management of Donors with Confirmed Positive Microbiological Markers, MPD/MED/009/05), but has never been evaluated in a systematic study. Worldwide, only a handful of studies have approached the issue (Tynell et al, 2007; Kleinman et al, 2004), but have suggested that donors can experience confusion and anxiety as a result of notification. It is therefore possible that current notification procedures do not adequately address the donors' needs.

A recent in-depth qualitative study of the impact of notification of possible increased risk of variant Creutzfeldt-Jacob Disease (vCJD) for public health purposes (Elam et al, awaiting publication) found that notification was a shocking event in most subjects' lives, although it did not have a lasting emotional impact. Several factors influenced how well information given at notification was retained and implemented. As it is anticipated that all blood donations are to be screened for vCJD as soon as a test becomes available, the need for the development of optimal notification procedures was identified. The proposed study builds on those findings.

Blood donors comprise a unique population, usually characterised by high altruism, low risk-taking, conservatism and concern with health (Simmons et al., 1993; Burnett, 1981). For those reasons, notification of serious infection could cause them greater distress, experience of stigma and self-image damage than an average person (Jackson, 2005; Orsini, 2002; Schulte, 2002; Murray, 1990), and therefore should be handled with utmost care.

Currently, blood donations in the UK are routinely tested for syphilis, hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) and human T-lymphotropic virus (HTLV). Additionally, if indicated by donor history, supplementary tests for malaria, T-cruzi, cytomegalovirus (CMV), and West Nile virus (WNV) are performed. For the purposes of the study, only donors notified of positive test results of routine screening will be surveyed. Those testing positive for syphilis will not be included because of the universally curable nature of the infection.

A mail out questionnaire was chosen as the best form of data collection because of the significant dispersion of the study population, the continuity of contact method, and the low intrusiveness of the instrument. Those wishing to participate will be able to complete the questionnaire at a time and place most convenient to them. As initial communication was by letter, it is expected that a mail out survey accompanied by a cover letter will be accessible to most donors. A telephone- and a web-based survey completion option will also be offered to facilitate access.

The questionnaire will focus on three main areas of interest, namely satisfaction, emotional response and understanding. These were identified from the in-depth vCJD study, donor records and literature review as the issues most pertinent to the notification process, and ones influenced by the manner in which information is provided. Personal characteristics and circumstances will not be considered, as they are already well researched from the perspective of coping (Kaye & Raghavan, 2002; Baile et al., 2000; Kraus et al., 2000; Buckman & Kason, 1992), and not controlled for in blood donation, thus limiting their usefulness for informing donor notification process.

To ensure the appropriateness and feasibility of questions, and to avoid misrepresentation, the survey will be piloted with a small sample of donors testing positive in routine screening in 2007.

The return of a completed questionnaire will be treated as implied consent, and the return of an empty one with or without the opt-out option selected will be taken to signify the donor's decision not to give such consent.

The main risk identified in contacting positive donors is re-traumatisation, and a helpline number will be provided to allow those experiencing any distress to discuss their situation. It is hoped, however, that as the infections under study are chronic, re-traumatisation would be rare and minimal. It is further hoped that the character of the project, which aims to aid the development of notification procedures that would be the most satisfactory to donors receiving positive test results in the future, would be welcome by most subjects as an opportunity to engage in an activity that could be of benefit to others. Should any donor's reaction suggest that their situation may be serious, every attempt will be made to offer follow-up care. Any aggravating issues inherent in the questionnaire itself, however, will hopefully be identified and rectified at the piloting stage. The direct donor burden, should they choose to participate in the study, should be limited to the 20-30 minutes needed to complete the questionnaire.

Only the Principal Investigator and the researcher will have access to identifiable personal data, the PI as a member of the donor's healthcare team, and the researcher within the remit of the position. The researcher's access to and use of donor records will comply with the Good Clinical Practice guidelines, and further with the NHS Confidentiality Code of Practice. Donor name and number will be coded and stored separately from the pseudonymised survey data. The file linking donor identifiable information with codes will be stored for the duration of the research project only. The raw survey data file and returned questionnaires will be stored securely for a minimum of 2 years. Only the pseudonymised data will be used for analysis, and no identifiable donor information will be included in ensuing reports.

The demographic data such as age, ethnicity and sex already available in the donor records will be pseudonymised and used to reduce response burden. Only the data theoretically relevant to the study will be included. The access to all study files will be restricted, and all information will be stored and shared securely as per NHS guidelines. No identifiable personal data will be shared.

The survey data will be statistically analysed using SPSS. Every attempt will be made to assess the extent of the non-response error using pseudonymised demographic data of the non-respondents. Due to the large number of variables involved, main attention will be given to descriptive statistics.

To avoid misinterpretation, any conclusions drawn from the data will be discussed by the Project Management Group and not made by the researcher in isolation. The results of the study will be published and accessible to the participants and general public in this way, or if requested directly.

Both the PI and the researcher are the employees of the NHSBT. The proposed research project is funded by the four UK blood services, and aims to improve the service offered. It will consider all responses, and use them to the benefit of the service users; however, it is intended to investigate the responses of blood donors who have donated in England or North Wales only. Due to the unique characteristics of this group, without further study the results cannot be generalised to the entire UK population or to other countries.

ELIGIBILITY:
Inclusion Criteria:

* deferred blood donor status, and
* deferral due to a positive result of a routine blood test for HIV, or hepatitis B, or hepatitis C, or HTLV, or having been identified as at risk of vCJD; and
* deferral occured in 2008 or 2009 (2007 for the pilot; 2005 for those at risk of vCJD); and
* donor registered at one of the NHSBT centres (English Blood Service in England and Wales);

Exclusion Criteria:

* not a blood donor; or
* no record of notification having taken place; or
* a member of Armed Forces or other profession where contact at the address provided could lead to a breach of confidentiality; or
* deferred before 2008 (if not in the pilot or notified of increased risk of vCJD);
* deferred as a result of a non-routine test or syphilis infection only; or
* donor registered with and notified by the Welsh, Scottish or Northern Irish Blood Services;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All donors testing positive for microbiology markers in 2008 and 2009, and those identified as at risk of vCJD in 2008.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the study is the reported level of satisfaction with the notification process, including the information provided and the donor's emotional response. | July-August 2010

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Hewitt, FRCP FRCPath, Principal Investigator — NHS Blood and Transplant; Theresa M Marteau, PhD FMedSci, Study Director — King's College London; Cameron F Ousbey, MSc, Study Director — NHS Blood and Transplant
Locations (1):
- NHS Blood and Transplant, Transfusion Microbiology, Colindale, London, United Kingdom

REFERENCES:
- [Background] Elam G, Oakley K, Connor N, Hewitt P, Ward HJ, Zaman SM, Chow Y, Marteau TM. Impact of being placed at risk of Creutzfeldt-Jakob disease: a qualitative study of blood donors to variant CJD cases and patients potentially surgically exposed to CJD. Neuroepidemiology. 2011;36(4):274-81. doi: 10.1159/000328646. Epub 2011 Jul 12. PMID 21757956
- [Background] French DP, Maissi E, Marteau TM. Psychological costs of inadequate cervical smear test results. Br J Cancer. 2004 Nov 29;91(11):1887-92. doi: 10.1038/sj.bjc.6602224. PMID 15534608
- [Background] Kleinman S, Wang B, Wu Y, Glynn SA, Williams A, Nass C, Ownby H, Busch MP; Retrovirus Epidemiology Donor Study. The donor notification process from the donor's perspective. Transfusion. 2004 May;44(5):658-66. doi: 10.1111/j.1537-2995.2004.03347.x. PMID 15104645
- [Background] Tynell E, Norda R, Ekermo B, Sanner M, Andersson S, Bjorkman A. False-reactive microbiologic screening test results in Swedish blood donors-how big is the problem? A survey among blood centers and deferred donors. Transfusion. 2007 Jan;47(1):80-9. doi: 10.1111/j.1537-2995.2007.01067.x. PMID 17207234
- [Result] Reynolds CA, Brailsford SR, Hewitt PE. Notifying blood donors of infection: results of a donor satisfaction survey. Transfus Med. 2015 Dec;25(6):358-65. doi: 10.1111/tme.12268. Epub 2015 Dec 28. PMID 26707828
- See also: WORLD HEALTH ORGANISATION, ca. 2009. Blood transfusion safety: Universal access to safe blood and blood products for transfusion. — http://www.who.int/bloodsafety/en/